CLINICAL TRIAL: NCT07078734
Title: Research Assistant
Brief Title: Acute Effects of Foam Roller and Mulligan Technique on Hamstring Flexibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Abdulkadir Ertürk, Research assistant, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Kdrertrkfoam
Record Dates: First submitted 2025-07-12; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Hamstring Shortness
Keywords: Hamstring Shortness; Foam roller; Mulligan straight leg raise technique

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foam roller group (Active Comparator): The foam roller group is the group where the person uses his/her own weight to swing the hamstring muscle with a foam roller.
  Interventions: Other: Foam roller technique
- Mulligan Straight Leg Raise Technique (Active Comparator): This is a technique applied by a practitioner to this group of people with hamstring tightness.
  Interventions: Other: Mulligan Straight Leg Raise Technique

INTERVENTIONS:
Other: Foam roller technique — In this intervention group, the patient is given back and forth oscillations using his or her own weight using a foam roller under the supervision of a physiotherapist.
  Arms: Foam roller group
Other: Mulligan Straight Leg Raise Technique — This intervention consists of the mulligan straight leg raise technique applied to the patient by a physiotherapist.
  Arms: Mulligan Straight Leg Raise Technique

SUMMARY:
The hamstring muscle group is located at the back of the thigh. Due to its structure and people's habits, shortness in this muscle group is frequently observed. Shortness can cause problems such as low back pain, gait disturbances, thigh pain, and more. Numerous exercises and treatment methods have been used to restore flexibility to this muscle. This study will examine the acute effects of mulligan straight leg raises and foam rolling on university students with short hamstrings.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Hamstring tightness

Exclusion Criteria:

* Raise their legs straighter than 85-90 degrees
* Who have been actively engaged in regular sports for 2 years
* Who have had a lower extremity injury within the last 6 months
* Who have a neurological disease, or whose evaluation was incomplete for any reason.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
Active Knee Extension Test | day 1
  The individual is asked to actively extend the knee while the hip and knee are in a 90˚ flexion position.
Sit and Reach Test: | day 1
  Participants remove their shoes, place the soles of their feet on the sit-and-reach box, and, without bending their knees, reach forward as far as possible by placing their hands on top of each other. The distance between them is measured.
Knee Flexion-Extension Joint Range of Motion | day 1
  It refers to the participants' knee extension and flexion joint range of motion. It is measured with a goniometer by the physiotherapist after the appropriate position is given.

SECONDARY OUTCOMES:
Y Balance Test | day 1
  The subject is asked to stand with one foot in the middle and extend as far as possible along a Y line, which is 135˚ between the anterior and posterior directions and 90˚ between the posteromedial and posterolateral directions. The starting distance and the final distance are measured.
Hamstring and quadriceps muscle strenght | day 1
  This test evaluates hamstring and quadriceps muscle strength. Muscle strength will be measured using the Power Track 2 Commender device after the physiotherapist has instructed participants in the necessary measurement positions.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma ÜNVER, Professor, Study Director — Pamukkale University Faculty of Health Sciences
Locations (1):
- Pamukkale University Physical Therapy and Rehabilitation Faculty, Denizli, Pamukkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No